CLINICAL TRIAL: NCT03540940
Title: The Effect of Positive End-expiratory Pressure During Induction of General Anesthesia on Atelectasis Formation and Non-hypoxic Apnea Time in Small Children: a Randomized Controlled Trials
Brief Title: PEEP During Induction of Anesthesia in Small Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H 1804-100-938
Record Dates: First submitted 2018-05-17; First posted 2018-05-30 (Actual); Last update posted 2019-08-19 (Actual); Status verified 2019-08

CONDITIONS: Pediatric Anesthesia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- zero positive end expiratory pressure (Experimental)
  Interventions: Other: ZEEP
- Positive end expiratory pressure (Experimental)
  Interventions: Other: PEEP

INTERVENTIONS:
Other: PEEP — 7cmH2O positive end expiratory pressure
  Arms: Positive end expiratory pressure
Other: ZEEP — 0 cmH2O positive end expiratory pressure
  Arms: zero positive end expiratory pressure

SUMMARY:
Positive end-expiratory pressure (PEEP) applied during induction of anesthesia prevents atelectasis formation and increases the duration of nonhypoxic apnea in obese and nonobese patients. PEEP also prevents atelectasis formation in pediatric patients. Because pediatric patients arterial desaturation during induction of anesthesia develops rapidly, we studied the clinical benefit of PEEP applied during anesthesia induction.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients undergoing general anesthesia using endotracheal intubation

Exclusion Criteria:

* previous history of lung disease
* anticipated difficulty in airway management

Ages: 1 Month to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-05-21 (Actual); Primary Completion 2019-08-14 (Actual); Study Completion 2019-08-14 (Actual)

PRIMARY OUTCOMES:
Duration of Apnea | from the start of apnea until SpO2 reached 95%, maximum 5 minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, Professor, Principal Investigator — Seoul National University Hospital
Locations (2):
- South Korea (2):
  - Hee-Soo Kim, Seoul, Soul-t'ukpyolsi
  - Seoul National University Hospital, Seoul

REFERENCES:
- [Derived] Kim EH, Lee JH, Jang YE, Ji SH, Cho SA, Kim JT, Kim HS. Effect of positive end-expiratory pressure during anaesthesia induction on non-hypoxic apnoea time in infants: A randomised controlled trial. Eur J Anaesthesiol. 2021 Oct 1;38(10):1012-1018. doi: 10.1097/EJA.0000000000001400. PMID 33259454